CLINICAL TRIAL: NCT02522819
Title: Feasibility Evaluation of Continuous Positive Airway Pressure (CPAP) in the Treatment of Obstructive Sleep Apnea Synchrone in the Acute Phase of Stroke
Brief Title: Feasibility Evaluation of CPAP in the Treatment of Obstructive Sleep Apnea Synchrone in the Acute Phase of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1108101
Record Dates: First submitted 2015-08-12; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; acute stroke; apnea-hypopnea index (AHI)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- obstructive sleep apnea in the acute phase of stroke (Experimental): Use of CPAP over 5 nights for the treatment of obstructive sleep apnea in the acute phase of stroke
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Use of CPAP over 5 nights for the treatment of obstructive sleep apnea in the acute phase of stroke.

SUMMARY:
This project is focused on the treatment of obstructive sleep apnea in the acute phase of stroke. Stroke is a frequent pathology with a high morbidity and mortality rate. Although it has now been proved that obstructive sleep apnea syndrome (OSAS) is a risk factor of stroke, on the other hand, there is evidence that 50 to 70% of patients in the acute phase of stroke have obstructive sleep apnea (OSA) based on an apnea-hypopnea index (AHI) of ≥ 10. OSA is associated with worse functional outcomes and higher mortality in the post-stroke period. Profound hemodynamic fluctuations and hypoxia generated by sleep apnea are likely to aggravate cerebral ischemia, particularly in the acute phase of stroke in the potentially reversible ischemic penumbra. Continuous Positive Airway Pressure (CPAP) is the primary treatment for obstructive sleep apnea.

Yet, to our knowledge, there have been very few studies aimed at demonstrating the value of CPAP in the treatment of obstructive sleep apnea in the acute phase of stroke. Only one randomised trial has provided the means to document neurological improvement at mid term (1 month) in a targeted population.

Before undertaking a comparative study evaluating the efficacy of CPAP in the acute phase of ischemic stroke, it is worth evaluating the feasibility and tolerance of introducing CPAP at the very early stage of ischemic stroke. Therefore, the purpose of our study is to evaluate the feasibility of CPAP in the treatment of OSA in the acute phase of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* - Clinical presentation of ischemic stroke confirmed by imaging (CT or MRI brain scan)
* less than 24 hours from onset of symptoms
* admitted to the Neurovascular unit of the Emergency Hospitalisation Department of 'Hôpital Nord' of the university hospital of Saint-Étienne
* presenting obstructive sleep apnea syndrome (defined as an apnea-hypopnea index (AHI) of ≥ 10 and > 50% of obstructive events)
* written consent of patient

Exclusion Criteria:

* Concussion (Coma Glasgow Score <12)
* Comprehension aphasia
* Uncontrollable confusion and agitation
* History of dementia
* History of ischemic stroke with neurological damage
* History of hemorrhagic stroke
* History of epilepsy
* Cerebrospinal fluid leak, recent cranial surgery or head injury
* Serious bullous lung disease
* Hypoxic pulmonary disease
* Pleurisy or pneumothorax requiring draining
* Respiratory distress requiring mechanical ventilation
* Oxygen therapy prior to stroke
* Non-invasive ventilation therapy prior to stroke
* Hypotension
* Dehydration
* Hypersalivation
* Vomiting
* Pregnancy, parturients, breast feeding
* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
CPAP feasibility | day 5
  Number of patients for which CPAP is used for a minimum of 3 hours per night over 5 nights. CPAP feasibility is retained if at least 50% of all patients have had the use of CPAP for at least 3 hours per night over 5 nights.

SECONDARY OUTCOMES:
Feasibility of the ventilatory polygraph | night 1
  Number of readable polygraph recordings. A readable recording is defined as a minimum duration of 6 hours of recording with signals of a sufficient quality.
Tolerance of CPAP by patient per night | 5 nights
  Evaluation of CPAP tolerance according to a score as per the VAS (Visual Analogue Scale) for pain ranging from 0: "No tolerance" to 10: "Excellent tolerance" per night of use of CPAP device
Number of hypotensive episodes per night per patient | 5 nights
  Number of hypotensive episodes per night per patient by non-invasive measuring of blood pressure during the period of use of the CPAP device and defined according to systolic BP of < 90 mm Hg or drop of 40 mmHg with respect to the basic parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard TARDY, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France